CLINICAL TRIAL: NCT04550156
Title: Evaluation of the Introduction of a Colorectal Bundle in Left Sided Colorectal Resections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Hospital Centre Biel/Bienne (Other); Luzerner Kantonsspital (Other); Kantonsspital Aarau (Other); Kantonsspital Liestal (Other); Spital Limmattal Schlieren (Other); Kantonsspital Olten (Other); Clarunis - Universitäres Bauchzentrum Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EvaCol
Record Dates: First submitted 2020-08-19; First posted 2020-09-16 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Disorders; Surgery--Complications; Colorectal Cancer; Anastomotic Leak; Complication of Surgical Procedure
MeSH Terms: conditions — Colorectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, multicenter trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (No Intervention): Patients are treated according to current local standards
- Colorectal Bundle Arm (Experimental): Patients are treated according to the colorectal bundle
  Interventions: Procedure: Colorectal Bundle

INTERVENTIONS:
Procedure: Colorectal Bundle — 1. Preoperative optimization of the nutritional status: Perform nutritional risk screening (NRS), measure albumin or prealbumin preoperatively and initiate nutritional support
  2. Preoperative showering with an antiseptic agent
  3. Administer preoperative antibiotic prophylaxis
  4. Hair removal in the operative field with clippers
  5. Peri-, intra-, and postoperative warming to maintain body temperature
  6. Peri- and intraoperative glucose control
  7. Usage of a wound protection device
  8. Change of gloves and instruments after anastomosis
  9. Anastomosis only with experienced senior surgeon present in theatre for any elective and emergency procedures
  Arms: Colorectal Bundle Arm

SUMMARY:
The complication rate in colorectal surgery is high and shows a large variance depending on the patient and the treating surgeon. The primary aim of the presented study is to evaluate the introduction of a colorectal bundle to reduce the complication rate in left sided colorectal resections. The colorectal bundle is a catalog of measures consisting of several items These are for example preoperative risk stratification, antibiotic and mechanical bowel preparation and preoperative showering. The primary endpoint will be the complication rate measured as the comprehensive clinical index (CCI) within 30 days. Investigators will include patients that undergo elective or emergency left sided colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 years
* Patients undergoing any left sided emergency or elective colorectal resections
* Patients should have given or will give a general consent

Exclusion Criteria:

* no general consent given
* unable to provide informed general consent
* vulnerable patients (Age < 18 years or patients with severe dementia)
* the intervention is a reoperation within 30 days of primary operation

Exclusion criteria for an antibiotic decontamination subgroup:

* known allergy to one of the applied antibiotic regimes
* active bacterial infection requiring systemic antibiotics
* IV or oral antibiotics in past 7 days prior to the planned decontamination
* terminal kidney disease
* unable to take antibiotic decontamination medication
* pregnancy or breastfeeding
* emergency or expedited surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1141 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Comprehensive complication index | 30 days
  The primary endpoint is the comprehensive complication index (CCI) at 30 days after the index procedure, a continuous scale to measure surgical morbidity that has been developed on the basis of the Clavien Dindo Classification for surgical complications and summarizes and weighs all postoperative complications to a scale from 0 (no complications) to 100 (death of the patient) .

SECONDARY OUTCOMES:
Surgical side infections | 30 days
  Rate of surgical side infections within 30 days
Number of patients who died within 30 days | 30 days
  Postoperative mortality within 30 days
Hospital length of stay | immediately after discharge
  Length of hospital stay in days
Contribution margin | immediately after discharge
  Measured as the difference between allocated costs and billed and payed income for a particular case
Rate of anastomotic leakage | 30 days
  Any radiologically or clinically diagnosed anastomotic leakage

CONTACTS AND LOCATIONS:
Overall Officials: Marco von Strauss und Tourney, PD Dr., Principal Investigator — Clarunis - Universitäres Bauchzentrum Basel; Markus Zuber, Prof. Dr., Study Director — Clarunis - Universitäres Bauchzentrum Basel
Locations (7):
- Switzerland (7):
  - Kantonsspital Baselland, Liestal, Basel-Landschaft
  - Lantonsspital Aarau, Aarau, Canton of Aargau
  - Clarunis-universitäres Bauchzentrum, Basel, Canton of Basel-City
  - Spitalzentrum Biel, Biel/Bienne, Canton of Bern
  - Kantonsspital Luzern, Lucerne, Canton of Lucerne
  - Kantonsspital Olten, Olten, Canton of Solothurn
  - Spital Limmattal, Schlieren, Canton of Zurich

REFERENCES:
- [Background] Bergvall M, Skullman S, Kodeda K, Larsson PA. Better survival for patients with colon cancer operated on by specialized colorectal surgeons - a nationwide population-based study in Sweden 2007-2010. Colorectal Dis. 2019 Dec;21(12):1379-1386. doi: 10.1111/codi.14760. Epub 2019 Jul 30. PMID 31293019
- [Background] 2017 European Society of Coloproctology (ESCP) collaborating group. Safety of primary anastomosis following emergency left sided colorectal resection: an international, multi-centre prospective audit. Colorectal Dis. 2018 Sep;20 Suppl 6:47-57. doi: 10.1111/codi.14373. PMID 30255647
- [Background] 2017 European Society of Coloproctology (ESCP) Collaborating Group. The 2017 European Society of Coloproctology (ESCP) international snapshot audit of left colon, sigmoid and rectal resections - Executive Summary. Colorectal Dis. 2018 Sep;20 Suppl 6:13-14. doi: 10.1111/codi.14391. No abstract available. PMID 30255645
- [Background] Borstlap WAA, Westerduin E, Aukema TS, Bemelman WA, Tanis PJ; Dutch Snapshot Research Group. Anastomotic Leakage and Chronic Presacral Sinus Formation After Low Anterior Resection: Results From a Large Cross-sectional Study. Ann Surg. 2017 Nov;266(5):870-877. doi: 10.1097/SLA.0000000000002429. PMID 28746154
- [Background] Frasson M, Flor-Lorente B, Rodriguez JL, Granero-Castro P, Hervas D, Alvarez Rico MA, Brao MJ, Sanchez Gonzalez JM, Garcia-Granero E; ANACO Study Group. Risk Factors for Anastomotic Leak After Colon Resection for Cancer: Multivariate Analysis and Nomogram From a Multicentric, Prospective, National Study With 3193 Patients. Ann Surg. 2015 Aug;262(2):321-30. doi: 10.1097/SLA.0000000000000973. PMID 25361221
- [Background] Amri R, Dinaux AM, Kunitake H, Bordeianou LG, Berger DL. Risk Stratification for Surgical Site Infections in Colon Cancer. JAMA Surg. 2017 Jul 1;152(7):686-690. doi: 10.1001/jamasurg.2017.0505. PMID 28403477
- [Background] Bisig B, Gutzwiller F, Domenighetti G. [Incidence of operations in Switzerland related to insurance status]. Swiss Surg. 1998;4(3):109-16; discussion 116-7. German. PMID 9655004
- [Background] Haynes AB, Weiser TG, Berry WR, Lipsitz SR, Breizat AH, Dellinger EP, Herbosa T, Joseph S, Kibatala PL, Lapitan MC, Merry AF, Moorthy K, Reznick RK, Taylor B, Gawande AA; Safe Surgery Saves Lives Study Group. A surgical safety checklist to reduce morbidity and mortality in a global population. N Engl J Med. 2009 Jan 29;360(5):491-9. doi: 10.1056/NEJMsa0810119. Epub 2009 Jan 14. PMID 19144931
- [Background] Haugen AS, Softeland E, Almeland SK, Sevdalis N, Vonen B, Eide GE, Nortvedt MW, Harthug S. Effect of the World Health Organization checklist on patient outcomes: a stepped wedge cluster randomized controlled trial. Ann Surg. 2015 May;261(5):821-8. doi: 10.1097/SLA.0000000000000716. PMID 24824415
- [Background] Tanner J, Padley W, Assadian O, Leaper D, Kiernan M, Edmiston C. Do surgical care bundles reduce the risk of surgical site infections in patients undergoing colorectal surgery? A systematic review and cohort meta-analysis of 8,515 patients. Surgery. 2015 Jul;158(1):66-77. doi: 10.1016/j.surg.2015.03.009. Epub 2015 Apr 25. PMID 25920911
- [Background] Berrios-Torres SI, Umscheid CA, Bratzler DW, Leas B, Stone EC, Kelz RR, Reinke CE, Morgan S, Solomkin JS, Mazuski JE, Dellinger EP, Itani KMF, Berbari EF, Segreti J, Parvizi J, Blanchard J, Allen G, Kluytmans JAJW, Donlan R, Schecter WP; Healthcare Infection Control Practices Advisory Committee. Centers for Disease Control and Prevention Guideline for the Prevention of Surgical Site Infection, 2017. JAMA Surg. 2017 Aug 1;152(8):784-791. doi: 10.1001/jamasurg.2017.0904. PMID 28467526
- [Background] Fry DE. Review of The American Society of Colon and Rectal Surgeons Clinical Practice Guidelines for the Use of Bowel Preparation in Elective Colon and Rectal Surgery. JAMA Surg. 2020 Jan 1;155(1):80-81. doi: 10.1001/jamasurg.2019.4551. No abstract available. PMID 31693066
- [Background] McDermott FD, Heeney A, Kelly ME, Steele RJ, Carlson GL, Winter DC. Systematic review of preoperative, intraoperative and postoperative risk factors for colorectal anastomotic leaks. Br J Surg. 2015 Apr;102(5):462-79. doi: 10.1002/bjs.9697. Epub 2015 Feb 19. PMID 25703524
- [Background] Allegranzi B, Zayed B, Bischoff P, Kubilay NZ, de Jonge S, de Vries F, Gomes SM, Gans S, Wallert ED, Wu X, Abbas M, Boermeester MA, Dellinger EP, Egger M, Gastmeier P, Guirao X, Ren J, Pittet D, Solomkin JS; WHO Guidelines Development Group. New WHO recommendations on intraoperative and postoperative measures for surgical site infection prevention: an evidence-based global perspective. Lancet Infect Dis. 2016 Dec;16(12):e288-e303. doi: 10.1016/S1473-3099(16)30402-9. Epub 2016 Nov 2. PMID 27816414
- [Background] Bertschi D, Weber WP, Zeindler J, Stekhoven D, Mechera R, Salm L, Kralijevic M, Soysal SD, von Strauss M, Mujagic E, Marti WR. Antimicrobial Prophylaxis Redosing Reduces Surgical Site Infection Risk in Prolonged Duration Surgery Irrespective of Its Timing. World J Surg. 2019 Oct;43(10):2420-2425. doi: 10.1007/s00268-019-05075-y. PMID 31292675
- [Background] Hoang SC, Klipfel AA, Roth LA, Vrees M, Schechter S, Shah N. Colon and rectal surgery surgical site infection reduction bundle: To improve is to change. Am J Surg. 2019 Jan;217(1):40-45. doi: 10.1016/j.amjsurg.2018.07.008. Epub 2018 Jul 9. PMID 30025846
- [Background] Madrid E, Urrutia G, Roque i Figuls M, Pardo-Hernandez H, Campos JM, Paniagua P, Maestre L, Alonso-Coello P. Active body surface warming systems for preventing complications caused by inadvertent perioperative hypothermia in adults. Cochrane Database Syst Rev. 2016 Apr 21;4(4):CD009016. doi: 10.1002/14651858.CD009016.pub2. PMID 27098439
- [Background] de Vries FE, Gans SL, Solomkin JS, Allegranzi B, Egger M, Dellinger EP, Boermeester MA. Meta-analysis of lower perioperative blood glucose target levels for reduction of surgical-site infection. Br J Surg. 2017 Jan;104(2):e95-e105. doi: 10.1002/bjs.10424. Epub 2016 Nov 30. PMID 27901264
- [Background] Tanner J, Norrie P, Melen K. Preoperative hair removal to reduce surgical site infection. Cochrane Database Syst Rev. 2011 Nov 9;(11):CD004122. doi: 10.1002/14651858.CD004122.pub4. PMID 22071812
- [Background] Zhang L, Elsolh B, Patel SV. Wound protectors in reducing surgical site infections in lower gastrointestinal surgery: an updated meta-analysis. Surg Endosc. 2018 Mar;32(3):1111-1122. doi: 10.1007/s00464-017-6012-0. Epub 2017 Dec 27. PMID 29282577
- [Background] Junker T, Mujagic E, Hoffmann H, Rosenthal R, Misteli H, Zwahlen M, Oertli D, Tschudin-Sutter S, Widmer AF, Marti WR, Weber WP. Prevention and control of surgical site infections: review of the Basel Cohort Study. Swiss Med Wkly. 2012 Sep 4;142:w13616. doi: 10.4414/smw.2012.13616. eCollection 2012. PMID 22949137
- [Background] Boyce SA, Bartolo DC, Paterson HM; Edinburgh Coloproctology Unit. Subspecialist emergency management of diverticulitis is associated with reduced mortality and fewer stomas. Colorectal Dis. 2013 Apr;15(4):442-7. doi: 10.1111/codi.12022. PMID 22966859
- [Background] Slankamenac K, Graf R, Barkun J, Puhan MA, Clavien PA. The comprehensive complication index: a novel continuous scale to measure surgical morbidity. Ann Surg. 2013 Jul;258(1):1-7. doi: 10.1097/SLA.0b013e318296c732. PMID 23728278
- [Background] Rasmussen HH, Holst M, Kondrup J. Measuring nutritional risk in hospitals. Clin Epidemiol. 2010 Oct 21;2:209-16. doi: 10.2147/CLEP.S11265. PMID 21042553
- [Background] Hanley JA. Simple and multiple linear regression: sample size considerations. J Clin Epidemiol. 2016 Nov;79:112-119. doi: 10.1016/j.jclinepi.2016.05.014. Epub 2016 Jul 5. PMID 27393156
- [Derived] Wiesler B, Gass JM, Galli R, Worni M, Nebiker C, Muller A, Pabst M, Stimpfle D, Werlen L, von Strauss Und Torney M; Clarunis EvaCol Study Group. Is There Still a Need to Discuss the Use of Antibiotic Decontamination? Results of a Prospective Cohort Study Involving 999 Left-Sided Colorectal Resections. J Am Coll Surg. 2025 Sep 1;241(3):474-483. doi: 10.1097/XCS.0000000000001396. Epub 2025 Aug 14. PMID 40167266
- [Derived] Wiesler B, Gass JM, Viehl CT, Muller A, Metzger J, Hartel M, Nebiker C, Rosenberg R, Galli R, Zingg U, Ochsner A, Eisner L, Pabst M, Worni M, Henschel M, von Flue M, Zuber M, von Strauss Und Torney M. Evaluation of the Introduction of a Colorectal Bundle in Left Sided Colorectal Resections (EvaCol): Study Protocol of a Multicentre, Observational Trial. Int J Surg Protoc. 2022 Jul 14;26(1):57-67. doi: 10.29337/ijsp.177. eCollection 2022. PMID 35891921